CLINICAL TRIAL: NCT06345313
Title: The Effects of Surgery Performed At Different Times of the Day on Inflammation and Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Inflammation
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Inflammatory Response
Keywords: CIRCADIAN RHYTHM; POSTOPERATİVE RECOVERY

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Day Group (Active Comparator): Participants who underwent inguinal herniography operation between 08.00-12.00
  Interventions: Procedure: Day Group
- Night Group (Active Comparator): Participants who underwent inguinal herniography operation between 18.00-22.00
  Interventions: Procedure: Night Group

INTERVENTIONS:
Procedure: Day Group — Patient group that will be operated on between 08.00-12.00
  Arms: Day Group
Procedure: Night Group — Patient group that will be operated on between 18.00-22.00
  Arms: Night Group

SUMMARY:
To evaluate the inflammatory response of participants who will undergo unilateral inguinal hernia surgery at two different times of the day (08.00-12.00 during the day and 18.00-22.00 at night). The main question it aims to answer is; Is the inflammation response higher in participants who undergo surgery later in the day? Serum inflammatory parameters will be measured in both groups at the preoperative 1st hour and the postoperative 24th hour.

DETAILED DESCRIPTION:
Participants who would undergo unilateral inguinal herniography surgery at different times during the day were determined into two groups: day (08.00-12.00) and night (18.00-22.00). The Athens Insomnia Scale (AIS) will be asked verbally on the first preoperative day to determine the participants' preoperative circadian rhythm adaptation and sleep status. Serum inflammatory parameters of both participant groups will be measured and recorded at the preoperative 1st hour and the postoperative 24th hour. A laryngeal mask will be applied to the participants after induction with 2-3 mg/kg propofol and 1mg/kg fentanyl, as in routine anesthesia practice. Anesthesia maintenance will be provided with sevoflurane and 0.05-0.2 mcg/kg/min remifentanil infusion. Participants' age, gender, weight, height, BMI (body mass index), comorbidities, medications used, surgeries, ASA (American society of anesthesiologists) scoring, preoperative AIS (Athens insomnia scale) score, and preoperative laboratory data will be recorded. At the same time, participants' postoperative hospital stay, resting and moving NRS (Numeric rating scale) scores at the 24th postoperative hour, and recovery quality (Qor-15 score) from anesthesia will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American society of anesthesiologists) 1-2 adult participants between the ages of 18-70 who will undergo unilateral inguinal herniorrhaphy surgery at the Republic of Turkey Ministry of Health Ankara City Hospital.

Exclusion Criteria:

* Do not want to participate in the study
* Younger than 18 or older than 70
* Scores 6 and above on the preoperative Athens Insomnia Scale.
* ASA (American society of anesthesiologists) scores of 3 or greater than 3
* Have contraindications to the use of anesthetic drugs
* BMI>30 kg/m^2
* Have bilateral herniorrhaphy surgery
* Complicated inguinal hernia (incarcerated, strangulated…)
* Pregnancy
* Emergency surgeries
* Laparoscopic surgeries
* Develop an unexpected intraoperative surgical complication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Change of IL6 (interleukin6) (ng/ml) | Postoperative 24th hour
  IL6 (one of the inflammatory parameters, compared to baseline according to circadian rhythm) is a validated parameter that shows the severity of inflammation and trauma that can be measured in serum. Change = (postoperative 24th hour - preoperative 1st hour) higher difference means more inflammatory response.

SECONDARY OUTCOMES:
Quality of recovery from anesthesia according to difference in circadian rhythm | Postoperative 24th hour
  The quality of recovery-15 (QoR-15) is a patient-reported outcome measurement measuring QoR after surgery and anesthesia. The scale is arbitrary and ranges from 0 to 150. Higher results mean better build quality.
Change of NLR ( Neutrophil/ Lymphocyte Ratio ) | Postoperative 24th hour
  NLR (one of the inflammatory parameters, compared to baseline according to circadian rhythm) is a validated parameter that shows the severity of inflammation that can be measured in serum. Change = (postoperative 24th hour - preoperative 1st hour) higher difference means more inflammatory response.
Change of PLR ( Platelet / Lymphocyte Ratio ) | Postoperative 24th hour
  PLR (one of the inflammatory parameters, compared to baseline according to circadian rhythm) is a validated parameter that shows the severity of inflammation that can be measured in serum. Change = (postoperative 24th hour - preoperative 1st hour) higher difference means more inflammatory response.
Change of SII (Systemic immune-inflammation index ) | Postoperative 24th hour
  SII (Neutrophil × Platelet/ Lymphocyte) (one of the inflammatory parameters, compared to baseline according to circadian rhythm) is a validated parameter that shows the severity of inflammation that can be measured in serum. Change = (postoperative 24th hour - preoperative 1st hour) higher difference means more inflammatory response.
Change of CRP (C Reactive Protein) (mg/dl) | Postoperative 24th hour
  CRP (one of the inflammatory parameters, compared to baseline according to circadian rhythm) is a validated parameter that shows the severity of inflammation that can be measured in serum. Change = (postoperative 24th hour - preoperative 1st hour) higher difference means more inflammatory response.
Change of Fibrinogen (mg) | Postoperative 24th hour
  Fibrinogen (one of the inflammatory parameters, compared to baseline according to circadian rhythm) is a validated parameter that shows the severity of inflammation that can be measured in serum. Change = (postoperative 24th hour - preoperative 1st hour) higher difference means more inflammatory response.
Change of Sedimentation (mm/hour) | Postoperative 24th hour
  Sedimentation (one of the inflammatory parameters, compared to baseline according to circadian rhythm) is a validated parameter that shows the severity of inflammation that can be measured in serum. Change = (postoperative 24th hour - preoperative 1st hour) higher difference means more inflammatory response.
Change of Procalcitonin (µg/l) | Postoperative 24th hour
  Procalcitonin (one of the inflammatory parameters, compared to baseline according to circadian rhythm) is a validated parameter that shows the severity of inflammation that can be measured in serum. Change = (postoperative 24th hour - preoperative 1st hour) higher difference means more inflammatory response.
Change of Ferritin (ml/ng) | Postoperative 24th hour
  Ferritin (one of the inflammatory parameters, compared to baseline according to circadian rhythm) is a validated parameter that shows the severity of inflammation that can be measured in serum. Change = (postoperative 24th hour - preoperative 1st hour) higher difference means more inflammatory response.

OTHER OUTCOMES:
Numeric Rating Scale (NRS) | Postoperative 24th hour
  NRS is a scale that uses 11 numbers (between 0 and 10) to measure pain intensity. 0: no pain 10: unbearable pain

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, CANKAYA, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No